CLINICAL TRIAL: NCT00811317
Title: Closed-loop Glucose Control for Automated Management of Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Massachusetts General Hospital (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Edward R. Damiano, Associate Professor of Biomedical Engineering, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007P-000101; H-27207; SPID#0813
Record Dates: First submitted 2008-05-29; First posted 2008-12-18 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; glucose; hyperglycemia; hypoglycemia; insulin; glucagon; counter-regulation; closed-loop; feedback; control; dual-infusion; subcutaneous; automated; artificial pancreas; intensive insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hyperglycemia; Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Closed-loop (Experimental): Type 1 diabetic subjects under closed-loop blood glucose control
  Interventions: Device: Closed-loop

INTERVENTIONS:
Device: Closed-loop — Computer algorithm developed by Firas El-Khatib and Edward Damiano at Boston University that controls sub-cutaneous infusion of insulin and glucagon to regulate blood glucose to target

SUMMARY:
We hypothesize that our integrated closed-loop glucose-control system can provide effective, tight, and safe blood glucose (BG) control in type 1 diabetes, thereby establishing the feasibility of closed-loop BG control.

DETAILED DESCRIPTION:
This study investigates the utility of an integrated closed-loop glucose-control system for regulating BG in type 1 diabetic subjects. The closed-loop system utilizes sub-cutaneous infusion or insulin and glucagon under the control of a computer algorithm. The only inputs to the algorithm are the subject weight and BG values measured every five minutes. Subjects will undergo up to three 27 hour GCRC admissions during which they will consume three standardized meals. Subject may participate in up to two closed-loop visits (with different insulin lispro pharmacokinetic parameter settings in the control algorithm) and some subjects will participate in open-loop visits. During the closed-loop admission BG will be controlled by the closed-loop system. During the open-loop visit subjects will regulate their own BG in the usual function using their insulin pumps. A small group of non-diabetic subjects will undergo a single 27 hour GCRC admission during which they will eat the same standardized meals. During all admission BG will be measured every 5 minutes and blood will be collected for measurement of insulin and glucagon levels every 10 minutes. During the closed-loop admission of diabetic subjects and the single admission of non-diabetic subjects, three commercially available continuous glucose monitoring devices will be worn. The data from these devices will later be compared to reference BG data.

ELIGIBILITY:
Inclusion Criteria (type 1 diabetic subjects):

* Age 18 years or older
* Clinical type 1 diabetes for at least five years
* Otherwise healthy (mild chronic disease allowed if well controlled)
* Diabetes managed using an insulin infusion pump
* Body mass index (BMI) between 20 and 31
* Total daily dose (TDD) of insulin ≤ 1 U/kg and ≤ 100 U/day
* Post-prandial C-peptide < 0.1 nmol/L at 90 minutes in a mixed meal (Sustacal) tolerance test by the DCCT method
* Hemoglobin A1c less than or equal to 8.5%
* Prescription medication regimen stable for at least 1 month

Inclusion Criteria (non-diabetic subjects):

* Age 18 years or older
* No personal history of diabetes, impaired fasting glucose, or impaired glucose tolerance
* No personal history of pancreatic disease
* Not taking medication that may affect glucose, insulin, or glucagon dynamics
* Otherwise healthy (mild chronic disease allowed if well controlled)
* Body mass index (BMI) between 20 and 31
* Normal 75 g oral glucose tolerance test (fasting, 1 hour, and 2 hour measurements)

Exclusion Criteria (all subjects):

* Unable to provide informed consent or are unable to comply with study procedures
* Current participation in another clinical trial
* Anemia (HCT or hemoglobin less than normal for sex)
* Elevated alanine aminotransferase (ALT > 3 fold above upper limit of normal)
* Untreated or inadequately treated hyperthyroidism or hypothyroidism (abnormal TSH or free T4)
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception
* Progressive or proliferative diabetic retinopathy (subjects with mild, non-proliferative background retinopathy or stable disease previously treated with photocoagulation are not excluded).
* Renal insufficiency (creatinine clearance estimated by Cockcroft-Gault equation of ≤ 50 ml/min)
* Any known history or symptoms of coronary artery disease.
* Abnormal EKG
* Congestive heart failure
* History of TIA or stroke within preceding 6 months
* Acute illness or exacerbation of chronic illness at the time of the study procedure
* Change in medication regimen in the 30 days prior to enrollment
* History of seizures
* History of pheochromocytoma
* Abnormal plasma fractionated metanephrines
* History of adrenal disease or tumor
* History of pancreatic tumor, including insulinoma
* History of impaired gastric motility or gastroparesis requiring pharmacological or surgical treatment
* Current alcohol abuse (> 3 drinks daily) or substance abuse (any use within the last 6 months of illegal drugs)
* Severe mental illness (schizophrenia, bipolar disease, inadequately treated depression, or any psychiatric hospitalization in the last year)
* Impaired cognition or altered mental status.
* Hypertension (blood pressure > 140/90) at the time of screening
* Use of medications that reduce gastric motility
* Electrically powered implants that might be susceptible to RF interference
* Use non-insulin injectable anti-diabetic medications, inhaled insulin, or oral anti-diabetic medications
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
* Established history of latex, adhesive, tape allergy, inadequate venous access, history of allergy to or intolerance of aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, M.D., Ph.D., Study Director — Massachusetts General Hospital; Edward Damiano, Ph.D., Principal Investigator — Boston University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] El-Khatib FH, Jiang J, Gerrity RG, Damiano ER. Pharmacodynamics and stability of subcutaneously infused glucagon in a type 1 diabetic Swine model in vivo. Diabetes Technol Ther. 2007 Apr;9(2):135-44. doi: 10.1089/dia.2006.0006. PMID 17425438
- [Background] El-Khatib FH, Jiang J, Damiano ER. Adaptive closed-loop control provides blood-glucose regulation using dual subcutaneous insulin and glucagon infusion in diabetic Swine. J Diabetes Sci Technol. 2007 Mar;1(2):181-92. doi: 10.1177/193229680700100208. PMID 19888405
- [Background] El-Khatib FH, Jiang J, Damiano ER. A feasibility study of bihormonal closed-loop blood glucose control using dual subcutaneous infusion of insulin and glucagon in ambulatory diabetic swine. J Diabetes Sci Technol. 2009 Jul 1;3(4):789-803. doi: 10.1177/193229680900300428. PMID 20144330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed-loop
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Average Blood Glucose Over the Closed-loop Control Period
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
mg/dl | 164 (17)

2. Secondary Outcome: Percentage of Time Spent Within 70-180 mg/dl
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
percentage of time | 61 (15)

3. Secondary Outcome: Peak Hyperglycemia Following Each Meal
Time Frame: After each of 3 meals
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
mg/dl
  Breakfast | 226.7 (26.6)
  Lunch | 256.7 (30.7)
  Dinner | 276.5 (33.8)

4. Secondary Outcome: Percentage of Time Spent in Hyperglycemia (BG> 180 mg/dl) After Meals
Time Frame: After each of 3 meals
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
percentage of time | 38 (9)

5. Secondary Outcome: Percentage of Peak Post-prandial Hyperglycemias < 180 mg/dl (ADA Target)
Time Frame: 24 hours
Measure: Number; unit: percentage of blood glucose measurements
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
percentage of blood glucose measurements
  Breakfast | 6
  Lunch | 0
  Dinner | 0

6. Secondary Outcome: Percentage of Time Spent With BG < 70 mg/dl
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
percentage of time | 0.35 (0.33)

7. Secondary Outcome: Number of Hypoglycemic Events
Description: This outcome captures the number of hypoglycemic events that occurred throughout the entire study
Time Frame: 24 hours
Measure: Number; unit: Number of events
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
Number of events | 2

8. Secondary Outcome: Nadir Blood Glucose Level for Each Hypoglycemic Event
Time Frame: 24 hours
Measure: Number; unit: mg/dl
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
mg/dl
  Event 1 of 2 | 66
  Event 2 of 2 | 68

9. Secondary Outcome: Percentage of Time Spent With BG > 180 mg/dl
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
percentage of time | 38 (2.9)

10. Secondary Outcome: Total Insulin Dose
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: u/kg
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
u/kg | 0.67 (0.34)

11. Secondary Outcome: Glucagon T-max
Description: Time to maximum peak glucagon concentration
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
minutes | 23 (9)

12. Secondary Outcome: Total Glucagon Dose
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
mcg/kg | 3.5 (2.8)

13. Secondary Outcome: Blood Glucagon Levels
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: microgram/kg
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
microgram/kg | 1.7 (0.36)

14. Secondary Outcome: Average Glucose and Glycemic Variability (MAGE) During Closed Loop Control in Diabetic Subjects Compared to the Comparable 24-hour Period the Day Prior to Admission as Measured by Navigator CGM Data
Time Frame: 24 hours
Population: Navigator CGM data from the day prior to admission was not obtained
Arm/Group | Closed-loop
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Carbohydrate Interventions
Time Frame: 24 hours
Measure: Number; unit: number of interventions
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
number of interventions | 0

16. Secondary Outcome: Number of Participants Achieving a Stable Glucose Response to Insulin Dosing
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
participants | 11

17. Secondary Outcome: Number of Participants Achieving a Stable Glucose Response to Insulin Dosing Around Idle Times Prior to Meals
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
participants | 11

18. Secondary Outcome: Accuracy of the Continuous Glucose Monitor (CGM) Using Blood Glucose Measurement as the Standard
Description: Measuring the mean absolute relative difference (MARD) between the blood glucose measurement and CGM glucose readings, on three different CGM devices: Dexcom, Guardian and Navigator
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percent absolute difference
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
percent absolute difference
  Navigator CGM | 9.94 (10.09)
  Dexcom CGM | 22.55 (20.75)
  Guardian CGM | 18.04 (15.46)

19. Secondary Outcome: Average Glucose and Glycemic Variability During Closed Loop Control in Diabetic Subjects Compared to the Comparable 24 Hour Period in Non-diabetic Subjects
Time Frame: 24 hours
Population: This outcome was not analyzed. There were no experiments in non-diabetic subjects that we were able to make a comparison with
Arm/Group | Closed-loop
Number analyzed (Participants) | 0

20. Secondary Outcome: Insulin and Glucagon Levels During the Closed-loop Admission as Compared to the Comparable 24 Hour Period During the Open Loop Admission of Diabetic Subjects
Time Frame: 24 hours
Population: This outcome was not analyzed. There were no open loop experiments in diabetic subjects that we were able to make a comparison with
Arm/Group | Closed-loop
Number analyzed (Participants) | 0

21. Secondary Outcome: Sensitivity for Hypo- and Hyperglycemia of the CGM Devices Using the BG Measurement as the Standard
Description: Mean absolute relative difference (MARD) of CGM and BG glucose readings in hypoglycemia (< 70 mg/dl) and hyperglycemia (>180 mg/dl) in three different CGM devices: Dexcom, Navigator and Guardian
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percent absolute difference
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
percent absolute difference
  Dexcom < 70 | 18.90 (11.85)
  Navigator < 70 | 18.64 (16.96)
  Guardian < 70 | 36.46 (23.60)
  Dexcom > 180 | 20.28 (15.34)
  Navigator > 180 | 9.41 (8.78)
  Guardian > 180 | 20.71 (16.95)

22. Secondary Outcome: Set Point Using CGM Data as the Input to the Controller for Future Studies
Description: The algorithm in the Bionic Pancreas must have a pre-specified target glucose it is trying to achieve in order to make dosing decisions. Using data from this study, investigators planned to determine what an appropriate glucose target should be for future studies.
Time Frame: 24 hours
Measure: Number; unit: mg/dl
Arm/Group | Closed-loop
Number analyzed (Participants) | 11
mg/dl | 100

23. Secondary Outcome: Insulin and Glucagon Levels During Closed Loop and Open Loop Admissions of Diabetic Subjects Compared to the Comparable 24 Hour Period During the Admission of Non-diabetic Subject
Time Frame: 24 hours
Population: as for outcome 19
Arm/Group | Closed-loop
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Closed-loop
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No